CLINICAL TRIAL: NCT05188261
Title: A Phase 1 Placebo-controlled Study of the Safety and Tolerability of Rectally Administered Single Ascending Doses of IW-3300 in Healthy Volunteers
Brief Title: A Study of Single Ascending Doses of IW-3300 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: C3300-101
Record Dates: First submitted 2021-12-17; First posted 2022-01-12 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigator and all other clinical research unit staff, sponsor study personnel, and the participant will remain blinded to individual participant treatment assignments throughout the study. Treatment assignments of individual participants will only be unblinded to a sponsor representative for regulatory reporting purposes or if warranted by emerging safety or tolerability issues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: 100 μg IW-3300 (Experimental): Dose 1: within the cohort, 6 participants receive active drug (IW-3300)
  Interventions: Drug: IW-3300
- Cohort 1: Placebo (Placebo Comparator): Within the cohort, 2 participants will receive the matching placebo dose
  Interventions: Drug: Placebo
- Cohort 2: 300 μg IW-3300 (Experimental): Dose 2: within the cohort, 6 participants receive active drug (IW-3300)
  Interventions: Drug: IW-3300
- Cohort 2: Placebo (Placebo Comparator): Within the cohort, 2 participants will receive the matching placebo dose
  Interventions: Drug: Placebo
- Cohort 3: 900 μg IW-3300 (Experimental): Dose 3: within the cohort, 6 participants receive active drug (IW-3300)
  Interventions: Drug: IW-3300
- Cohort 3: Placebo (Placebo Comparator): Within the cohort, 2 participants will receive the matching placebo dose
  Interventions: Drug: Placebo
- Cohort 4: 2500 μg IW-3300 (Experimental): Dose 4: within the cohort, 6 participants receive active drug (IW-3300)
  Interventions: Drug: IW-3300
- Cohort 4: Placebo (Placebo Comparator): Within the cohort, 2 participants will receive the matching placebo dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IW-3300 — A single dose of IW-3300 administered rectally (as a low-volume [20 mL] enema) following a fast of at least 6 hours.
  Arms: Cohort 1: 100 μg IW-3300; Cohort 2: 300 μg IW-3300; Cohort 3: 900 μg IW-3300; Cohort 4: 2500 μg IW-3300
Drug: Placebo — A single dose of placebo administered rectally (as a low-volume [20 mL] enema) following a fast of at least 6 hours.
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo

SUMMARY:
This is a first-in-human study to evaluate the safety and tolerability of single ascending doses of IW-3300. The study drug will be administered rectally as a low-volume (20 mL) enema. Study participants will be randomized in a 3:1 ratio to receive a single dose of IW-3300 or placebo. Up to 5 different doses of IW-3300 will be studied. Safety reviews will be conducted before proceeding to each higher dose.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, randomized, double-blind, placebo-controlled, single-ascending-dose study assessing the safety, tolerability, and pharmacokinetics (PK) of IW 3300 administered rectally as a low-volume enema in healthy adult volunteers. This first-in-human study will assess participants for safety, tolerability, and PK.

The study includes up to 6 treatments: placebo and up to 5 dose levels of IW-3300 which will be determined after safety reviews of previous cohorts.

This study will enroll a maximum of 40 participants (up to 5 cohorts of 8 participants each). The 8 participants within each cohort will be randomized in a double-blind manner to receive a single dose of IW-3300 (6 participants) or placebo (2 participants), administered rectally as a low-volume [20 mL] enema. Each cohort will progress through a Screening Period, Clinic Period, and Follow-up Period. Treatment duration will be 1 day. Participants will remain in the Phase 1 unit for approximately 24 hours after dosing and will be contacted by phone for follow-up approximately 2 weeks after dosing. Total participation will be 22 to 45 days, including the Screening, Clinic, and Follow-up Periods.

ELIGIBILITY:
Inclusion Criteria:

1. Males and female subjects of non-childbearing potential
2. Ages 18 to 60 years
3. Medically healthy with no clinically significant findings during medical evaluation including physical examination, 12-lead electrocardiogram (ECG), and clinical laboratory tests.
4. Normal bowel movement frequency of formed stool at baseline (≥3 per week and ≤3 per day; average Bristol stool form scale (BSFS) score of >2 and <6).
5. Body mass index (BMI) within the range 18.5 to 35.0 kg/m2 (inclusive) at the Screening Visit.
6. Male subjects and female partners are willing to use double-barrier method of contraception during the study.
7. If subject is ≥45 years of age, subject is compliant with colorectal cancer screening guidelines according to the American College of Gastroenterology (ACG) Clinical Guidelines: Colorectal Cancer Screening 2021.

Exclusion Criteria:

1. Evidence or history of clinically significant acute or chronic disease, or clinically significant illness within 30 days of the Screening Visit.
2. History of clinically significant hypersensitivity or allergies to any of the inactive ingredients contained in the active or placebo drug products.
3. History of any condition that would interfere with their ability to receive an enema, or has had difficulty receiving an enema in the past.
4. Recent history of anal fissure, anal abscess, complicated hemorrhoids, or presence or history of inflammatory bowel disease.
5. Used a prescription medication during the 14 days before Check-in
6. Used any over-the-counter medications, including laxatives, and herbal supplements during the 7 days before Check-in.
7. Received a licensed or investigational vaccine during the 30 days before Check-in or is planning to receive any vaccine during the study.
8. Recently received or donated blood products.
9. Undergone a surgical procedure during the 30 days before Check-in, other than minor dermatologic procedures, or has a history of surgery involving the GI tract or anal canal (with the exception of endoscopic procedures, appendectomy, and cholecystectomy).
10. Received any investigational drug during the 30 days or 5 half-lives of that investigational drug (whichever is longer) before the Screening Visit, or is planning to receive another investigational drug at any time during the study.
11. Abnormal laboratory tests or clinically significant findings on safety tests conducted at the Screening Visit or at Check-in.
12. Confirmed or suspected infection with COVID-19 at the Screening Visit or Check-in.
13. Positive serology for human immunodeficiency virus (HIV) 1, HIV 2, or hepatitis B surface antigen (HBsAg), or positive for anti-HIV 1, anti-HIV 2, or anti hepatitis C virus (HCV) antibodies at the Screening Visit.
14. History of alcohol or drug addiction during the year before the Screening Visit, or has a positive drug or alcohol screen at the Screening Visit or Check-in.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ironwood Study Chair, Study Director — Ironwood Pharmaceuticals
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to include up to 5 cohorts with 8 participants per cohort. Within each cohort, participants were randomized to receive a single dose of IW-3300 (6 participants) or placebo (2 participants). Doses to be evaluated were 100, 300, 900, and 2500 μg. An optional 5th cohort was planned to test an IW-3300 dose of ≤ 2500 μg. Based on a blinded review of safety and tolerability data from Cohort 1 through 4, the Dose Escalation Committee decided not to enroll the optional 5th Cohort.
Pre-assignment Details: As pre-specified by the statistical analysis plan, for the analyses reported herein, data from the 2 participants dosed with placebo in each of the 4 cohorts were pooled into a single placebo group (N=8).
Groups:
- Placebo: Participants received a single dose of placebo administered rectally (as a low-volume [20 mL] enema) following a fast of at least 6 hours.
- 100 μg IW-3300: Participants received a single dose of 100 μg IW-3300 administered rectally (as a low-volume [20 mL] enema) following a fast of at least 6 hours.
- 300 μg IW-3300: Participants received a single dose of 300 μg IW-3300 administered rectally (as a low-volume [20 mL] enema) following a fast of at least 6 hours.
- 900 μg IW-3300: Participants received a single dose of 900 μg IW-3300 administered rectally (as a low-volume [20 mL] enema) following a fast of at least 6 hours.
- 2500 μg IW-3300: Participants received a single dose of 2500 μg IW-3300 administered rectally (as a low-volume [20 mL] enema) following a fast of at least 6 hours.
Period: Overall Study
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300 | 900 μg IW-3300 | 2500 μg IW-3300
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300 | 900 μg IW-3300 | 2500 μg IW-3300 | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (12.64) | 29.8 (13.04) | 48.2 (11.30) | 39.7 (13.62) | 43.3 (13.76) | 39.7 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 2 | 7
  Male | 7 | 5 | 4 | 5 | 4 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 3 | 3 | 13
  Not Hispanic or Latino | 5 | 4 | 4 | 3 | 3 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 4 | 6 | 4 | 4 | 23
  Black or African American | 3 | 2 | 0 | 1 | 1 | 7
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Other, Not Specified | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a treatment-emergent AE (TEAE) if the AE started after initial study drug administration and within 1 day of the last dose of study drug.
Time Frame: From first dose of study drug through 24 hours post-Day 1 dose
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300 | 900 μg IW-3300 | 2500 μg IW-3300
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participants | 2 | 1 | 0 | 1 | 2

2. Primary Outcome: Number of Participants With Serious TEAEs
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; or other situations such as important medical events that may not be immediately life threatening or result in death or hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. An SAE was considered a treatment-emergent SAE (serious TEAE) if the SAE started after initial study drug administration and within 1 day of the last dose of study drug.
Time Frame: From first dose of study drug through 24 hours post-Day 1 dose
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300 | 900 μg IW-3300 | 2500 μg IW-3300
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 24 hours post-Day 1 dose
Description: An AE was considered a treatment-emergent AE (TEAE) if the AE started after initial study drug administration and within 1 day of the last dose of study drug.
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300 | 900 μg IW-3300 | 2500 μg IW-3300
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/8 | 1/6 | 0/6 | 1/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | 100 μg IW-3300 (N=6) | 300 μg IW-3300 (N=6) | 900 μg IW-3300 (N=6) | 2500 μg IW-3300 (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT05188261/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT05188261/SAP_001.pdf